CLINICAL TRIAL: NCT02219711
Title: A Phase 1/1b Study of MGCD516 in Patients With Advanced Solid Tumor Malignancies
Brief Title: Phase 1/1b Study of MGCD516 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 516-001
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Advanced Cancer
Keywords: MGCD516; MET; AXL; RET; TRK; NTRK; DDR2; KDR; VEGFR; PDGFRA; KIT; Tyrosine kinase inhibitor; NSCLC; Non-small cell lung cancer; Head and neck cancer; Renal cell carcinoma; Prostate cancer; Phase 1; CBL; Sitravatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Carcinoma, Renal Cell; Prostatic Neoplasms | interventions — sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGCD516 (Experimental): MGCD516 oral capsule, administered in escalating doses in Phase 1, beginning with daily dosing and exploring other regimens as necessary, in 21 or 28 days cycles
  Interventions: Drug: MGCD516

INTERVENTIONS:
Drug: MGCD516 — MGCD516 is a small molecule inhibitor of several closely related receptor tyrosine kinases. MGCD516 capsules will be taken with water.
  Other Names: Sitravatinib

SUMMARY:
MGCD516 is a receptor tyrosine kinase (RTK) inhibitor shown in preclinical models to inhibit a closely related spectrum of RTKs including MET, AXL, MER, and members of the VEGFR, PDGFR, DDR2, TRK and Eph families. In this study, MGCD516 is orally administered to patients with advanced solid tumor malignancies to evaluate its safety, pharmacokinetic, metabolism, pharmacodynamic and clinical activity profiles.

During the Phase 1 segment, the dose and regimen of MGCD516 will be assessed; during the Phase 1b segment, the clinical activity of MGCD516 will be evaluated in selected patient populations.

Patients anticipated to be enrolled in Phase 1b will be selected based upon having a tumor type, including but not limited to, non small cell lung cancer and head and neck cancer positive for specific activating MET, NTRK2, NTRK3, or DDR2 mutations, MET or KIT/PDGFRA/KDR gene amplification, selected gene rearrangements involving the MET, RET, AXL, NTRK1, or NTRK3 gene loci, or having loss of function mutations in the CBL gene. In addition patients with clear cell renal cell carcinoma refractory to angiogenesis inhibitors or metastatic prostate cancer with bone metastasis will be enrolled.

DETAILED DESCRIPTION:
During the Phase 1 segment, the dose and regimen of MGCD516 will be assessed.

During the Phase 1b segment, the clinical activity of MGCD516 will be evaluated in selected patient populations. Patients anticipated to be enrolled in Phase 1b will be selected based upon the following cancer diagnosis:

Non-small cell lung cancer with genetic alterations in MET, AXL, RET, TRK, DDR2, KDR, PDGFRA, KIT or CBL.

Head and neck squamous cell carcinoma with genetic alterations in MET.

Clear cell renal cell carcinoma refractory to angiogenesis inhibitors.

Metastatic prostate cancer with bone metastases.

Other cancer diagnosis having a selected genetic alteration in MGCD516 target RTKs.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable solid tumor malignancy
* Standard treatment is not available
* Adequate bone marrow and organ function

Exclusion Criteria:

* History of a significant cardiovascular illness
* Prolonged corrected QT (QTc) interval
* Left ventricular ejection fraction < 40%
* Symptomatic or uncontrolled brain metastases
* Other active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-08; Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Type of dose limiting adverse event | Up to 3 weeks on treatment
Area under the plasma concentration versus time curve (AUC) of MGCD516 | Up to 72 hours
Peak Plasma Concentration (Cmax) of MGCD516 | Up to 72 hours

SECONDARY OUTCOMES:
Kind of metabolites of MGCD516 in blood plasma | Up to 9 weeks on treatment
Concentration of selected marker proteins in blood plasma | Up to 9 weeks on treatment
  Proteins include VEGF A, soluble VEGF-R2 and soluble MET
Percent of patients having objective disease response to treatment | Up to 1 year on treatment
  Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chao, MD, Study Director — Mirati Therapeutics Inc.
Locations (43):
- United States (37):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Holy Cross Michael & Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Florida Cancer Affiliates, Ocala, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Oncology Hematology,, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University Center for Advanced Medicine, St Louis, Missouri
  - CHI Health St Francis, Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Oncology Hematology West PC, Nebraska Cancer Specialists, Omaha, Nebraska
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - St. Francis Cancer Center, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - The Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Blue Ridge Cancer Care, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - University of Wisconsin, Madison, Wisconsin
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Korea Veterans Health Service, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

REFERENCES:
- [Derived] Bazhenova L, Kim DW, Cho BC, Goel S, Heist R, Werner TL, Eaton KD, Wang JS, Pant S, Adkins DR, Blakely CM, Yan X, Neuteboom S, Christensen JG, Chao R, Bauer T. Sitravatinib in patients with solid tumors selected by molecular alterations: results from a Phase Ib study. Future Oncol. 2024 Dec;20(39):3213-3227. doi: 10.1080/14796694.2024.2418285. Epub 2024 Nov 8. PMID 39513224
- [Derived] Pant S, Cho BC, Kyriakopoulos CE, Spira A, Tannir N, Werner TL, Yan X, Neuteboom S, Chao R, Goel S. Targeting multiple receptor tyrosine kinases with sitravatinib: A Phase 1b study in advanced renal cell carcinoma and castrate-resistant prostate cancer. Invest New Drugs. 2024 Oct;42(5):547-558. doi: 10.1007/s10637-024-01465-9. Epub 2024 Aug 21. PMID 39168901
- [Derived] Bauer T, Cho BC, Heist R, Bazhenova L, Werner T, Goel S, Kim DW, Adkins D, Carvajal RD, Alva A, Eaton K, Wang J, Liu Y, Yan X, Christensen J, Neuteboom S, Chao R, Pant S. First-in-human phase 1/1b study to evaluate sitravatinib in patients with advanced solid tumors. Invest New Drugs. 2022 Oct;40(5):990-1000. doi: 10.1007/s10637-022-01274-y. Epub 2022 Jun 29. PMID 35767205